CLINICAL TRIAL: NCT06967155
Title: Non-randomised, Multicentre, Prospective, Single-arm, Phase II Study of the Efficacy and Toxicity of a Combination of Irinotecan With Dabrafenib and Trametinib, Anti-EGFR in the Second Line of Treatment of Patients With Metastatic BRAF V600E- Mutated Colorectal Cancer.
Brief Title: A Study of Irinotecan With Dabrafenib Plus Trametinib and Anti-EGFR in the Second Line of Therapy in People With Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Collaborators: City Clinical Oncology Hospital No 1 (Other Government); Moscow City Oncology Hospital No. 62 (Other Government); The Loginov MCSC MHD (Unknown); MMCC Kommunarka MHD (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05202500302
Record Dates: First submitted 2025-04-25; First posted 2025-05-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms
Keywords: metastatic colorectal cancer; BRAF V600E- mutated; treatment
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: * Drug: Dabrafenib
  * Drug: Trametinib
  * Drug: Cetuximab
  * Drug: Рanitumumab
  * Drug: Oxaliplatin
  * Drug: Irinotecan
  * Drug: Leucovorin
  * Drug: 5-FU
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan + Dabrafenib + Trametinib and Cetuximab or Panitumumab in the second line of therapy (Experimental): Irinotecan + Dabrafenib + Trametinib and Cetuximab or Panitumumab in the second line of therapy Dabrafenib 150 mg twice orally daily Trametinib 2 mg orally once daily Cetuximab 500 mg/m2 (120-minute IV infusion) every two weeks or Panitumumab 6 mg/kg (60-minute IV infusion) every two weeks Irinotecan 90 mg/m2 (90-minute IV infusion) weekly.
  Second-line treatment is administered until disease progression or intolerable toxicity. It may be possible to switch to a regimen of dabrafenib, trametinib, cetuximab or panitumumab if irinotecan is intolerable.
  Interventions: Drug: • Drug: Dabrafenib • Drug: Trametinib • Drug: Cetuximab • Drug: Рanitumumab • Drug: Oxaliplatin • Drug: Irinotecan • Drug: Leucovorin • Drug: 5-FU

INTERVENTIONS:
Drug: • Drug: Dabrafenib • Drug: Trametinib • Drug: Cetuximab • Drug: Рanitumumab • Drug: Oxaliplatin • Drug: Irinotecan • Drug: Leucovorin • Drug: 5-FU — Irinotecan + Dabrafenib + Trametinib and Cetuximab or Panitumumab in the second line of therapy Dabrafenib 150 mg twice orally daily Trametinib 2 mg orally once daily Cetuximab 500 mg/m2 (120-minute IV infusion) every two weeks or Panitumumab 6 mg/kg (60-minute IV infusion) every two weeks Irinotecan 90 mg/m2 (90-minute IV infusion) weekly.
  Second-line treatment is administered until disease progression or intolerable toxicity. It may be possible to switch to a regimen of dabrafenib, trametinib, cetuximab or panitumumab if irinotecan is intolerable.

SUMMARY:
The purpose of this study is to evaluate the efficacy and toxicity of irinotecan with dabrafenib, cetuximab/panitumumab in the second line of treatment for the potential treatment of colorectal cancer that: has a metastatic, inoperable; has a mutation in the BRAF gene.

Participants in this study will receive one of the following study treatments:

These participants will receive in the second line is irinotecan, dabrafenib + trametinib, cetuximab or panitumumab.

This trial is currently enrolling participants who will receive either irinotecan and dabrafenib plus cetuximab or panitumumab in the second line of therapy.

The study team will monitor how each participant responds to the study treatment for up to about 3 years.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the efficacy and toxicity of irinotecan in combination with dabrafenib + trametinib and cetuximab or panitumumab in second-line treatment of patients with metastatic inoperable colorectal cancer who have a BRAF mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic inoperable colorectal adenocarcinoma
2. The tumour has a BRAF mutation
3. Adequate function of hematopoiesis and basic indicators of internal organs
4. Has measurable or evaluable disease according to Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
5. Absence of grade 2 or higher toxicity from previous line of treatment.
6. It is possible to include patients with MSI or dMMR if they have received first-line immune checkpoint therapy.
7. ECOG PS 0-1

Exclusion Criteria:

1. Participants having more than 2 lines of treatment (a progression of disease within 12 months of the completion of adjuvant and/or perioperative chemotherapy with oxaliplatin and fluoropyrimidines is acceptable).
2. Presence of any other malignancy, except radically treated basal cell carcinoma, cervical cancer in situ, currently or within 5 years prior to enrolment.
3. Pregnant and breastfeeding women.
4. Male and female patients with preserved reproductive potential who refused to use adequate contraception throughout the study.
5. HIV-infected patients.
6. Patients with a life expectancy of less than 3 months.
7. The presence of a disease or condition that, in the opinion of the investigator, prevents the patient from participating in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-11-10 (Estimated); Study Completion 2028-06-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | assessed up to 12 months
  From date of enrollment until the date of first documented progression

SECONDARY OUTCOMES:
Progression-free survival | assessed up to 24 months
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first
Time to objective response | assessed up to 6 months
  Time from start of treatment to objective response to treatment
Duration of response | assessed up to 12 months
  Calculated from achieving objective response to progression or death from any cause
Disease control rate | Percentage of patients who achieved a complete response, partial response or disease stabilisation? through study completion, an average of 1 year
Overall survival | assessed up to 36 months
  From the time of enrolment until the death from any cause
Incidence of adverse events | Proportion of patients with adverse events out of all patients (NCI CTCAE 5.0)
Incidence of adverse events grade 3-4 | Proportion of patients with adverse events grade 3-4 out of all patients (NCI CTCAE 5.0)
Reduction of dose reductions and drug withdrawals | Proportion of patients with dose reductions and drug withdrawals in the total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Fedyanin MD, Principal Investigator — Blokhin's Russian Cancer Research Center
Locations (1):
- Blokhin's Russian Cancer Research Center, Moscow, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No